CLINICAL TRIAL: NCT01053702
Title: Study of the Safety and Efficacy of REGN475(SAR164877) in Patients With Pain Resulting From Thermal Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Medical Director, Regeneron Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R475-PN-0909
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Thermal Injury Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose 1 (Experimental): R475
  Interventions: Drug: R475
- Dose 2 (Experimental): R475
  Interventions: Drug: R475
- Dose 3 (Placebo Comparator): Placebo to match R475 dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: R475 — IV
  Arms: Dose 1; Dose 2
Drug: Placebo — Placebo
  Arms: Dose 3

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, single-dose study of the efficacy of REGN475 in patients with pain due to thermal injury.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ages 18 to 50, who have been hospitalized as a result of thermal injury
2. Moderate to severe procedural pain intensity (during wound care) on each of the initial assessment days

Exclusion Criteria:

1. Patients with burns caused by chemical exposure or electricity
2. Patients with inhalation injury or with evidence of pneumonia, cellulitis, or infection
3. Patients with traumatic musculoskeletal injuries (eg, bone fractures or dislocations) or traumatic head or chest injuries
4. Significant pre-injury concomitant illness such as, but not limited to, cardiac, renal, neurological, endocrinological, metabolic, psychiatric (including significant anxiety or depression), lymphatic disease, or drug dependence (alcohol or drug abuse), that would adversely affect the patient's management, recovery, or affect mortality or the patient's compliance with protocol assessments.
5. Women who are pregnant or nursing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in procedural pain intensity

SECONDARY OUTCOMES:
Cumulative analgesic usage
Weekly Patient-rated Global Impression of Change
Additional quality of life assessments

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tiseo, PhD, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Tampa, Florida, United States